CLINICAL TRIAL: NCT04355364
Title: Efficacy and Safety of Dornase Alfa Aerosol in ARDS Secondary to SARS-CoV-2 Coronavirus Respiratory Infection - COVID-19
Brief Title: Efficacy and Safety of aerosolizedDornase Alfa Administration in Patients With COVID19 Induced ARDS (COVIDORNASE)
Acronym: COVIDORNASE
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: No signal of benefit of treatment.
Sponsor: Fondation Ophtalmologique Adolphe de Rothschild (Network)
Collaborators: University Hospital, Strasbourg, France (Other); Centre Hospitalier Régional Metz-Thionville (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CGE_2020_9
Record Dates: First submitted 2020-04-15; First posted 2020-04-21 (Actual); Last update posted 2022-01-11 (Actual); Status verified 2021-12

CONDITIONS: COVID-19; Acute Respiratory Distress Syndrome
MeSH Terms: conditions — COVID-19; Respiratory Distress Syndrome | interventions — dornase alfa

STUDY DESIGN:
Intervention Model Description: Dornase alfa will be administered by nebulization, at a dose of 2500 IU twice daily, 12 hours apart, for 7 consecutive days, using a vibrating mesh nebulizer. The remainder of the management will be performed in accordance with good practice, including mechanical ventilation (protective ventilation, PEEP > 5 cmH2O, tracheal balloon pressure checking every 4 hours or automatic device, 30° head of the bed elevation, tidal volume 6-8mL/kg, plateau pressure < 30cmH2O), neuromuscular blockers if necessary, prone position if PaO2/FiO2<150, early enteral nutrition, glycemic control, a sedation protocol based on the RASS score.tracheal balloon pressure checking every 4 hours or automatic device, 30° head of the bed elevation, tidal volume 6-8mL/kg, plateau pressure < 30cmH2O), neuromuscular blockers if necessary, prone position if PaO2/FiO2<150, early enteral nutrition, glycemic control, a sedation protocol based on the RASS score.
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): Dornase alfa will be administered by nebulization, at a dose of 2500 IU twice daily, 12 hours apart, for 7 consecutive days, using a vibrating mesh nebulizer. The remainder of the management will be performed in accordance with good practice, including mechanical ventilation (protective ventilation, PEEP > 5 cmH2O, tracheal balloon pressure checking every 4 hours or automatic device, 30° head of the bed elevation, tidal volume 6-8mL/kg, plateau pressure < 30cmH2O), neuromuscular blockers if necessary, prone position if PaO2/FiO2<150, early enteral nutrition, glycemic control, a sedation protocol based on the RASS score.
  Interventions: Drug: Dornase Alfa Inhalation Solution [Pulmozyme]
- Control group (Active Comparator): Patients will receive the usual care in accordance with good practice.
  Interventions: Procedure: standard procedure

INTERVENTIONS:
Drug: Dornase Alfa Inhalation Solution [Pulmozyme] — Administered by nebulization, at a dose of 2500 IU twice daily, 12 hours apart, for 7 consecutive days
  Arms: Experimental group
Procedure: standard procedure — Patients will receive the usual care in accordance with good practice.
  Arms: Control group

SUMMARY:
This study plans to learn more about the effects of Dornase Alfa in COVID19 (coronavirus disease of 2019) patients, the medical condition caused by the Severe Acute Respiratory Syndrome Coronavirus 2 (SARS-CoV-2). Dornase Alfa is a FDA-approved drug for the treatment of cystic fibrosis, which facilitates mucus clearance by cutting apart neutrophil-derived extracellular double-stranded DNA. This study intends to define the impact of aerosolized intra-tracheal Dornase Alfa administration on the severity and progression of acute respiratory distress syndrome (ARDS) in COVID-19 patients. This drug might make lung mucus thinner and looser, promoting improved clearance of secretions and reduce extracellular double-stranded DNA-induced hyperinflammation in alveoli, preventing further damage to the lungs.

The study will recruit mechanically ventilated patients hospitalized in ICU who have been diagnosed with COVID-19 and meet ARDS criteria. It is a prospective, randomized, controlled, multicentric, open-label clinical trial.

The goal is to recruit 100 patients.

DETAILED DESCRIPTION:
Acute Respiratory Distress Syndrome (ARDS) is the most severe form of COVID-19 with a mortality reaching 50%. To date, no specific therapy has been shown to be effective. During an acute viral respiratory infection, lungs are the site of an intense neutrophil recruitment. Recruited neutrophils generate NETs (extracellular neutrophil traps) in the alveoli and bronchioles. NETs have been shown to be involved in bronchoalveolar congestion and amplification of the inflammatory response during viral pneumonia responsible for ARDS. Deoxyribonuclease 1 (DNAse 1) is an enzyme capable of cutting apart extracellular DNA strands, the backbone of NETs. The administration of recombinant human DNAse 1 (dornase alfa) leads to the loosening of the broncho-alveolar mucus and to a reduction in the inflammatory response within the alveoli.

By conducting a randomized, open-label, multicenter, controlled trial, our goal is to evaluate the efficacy and safety of aerosolized intra-tracheal dornase alfa administration in mechanically ventilated patients hospitalized for COVID19-related ARDS.

This is a randomized, controlled, multicentric, open-label clinical trial to evaluate the efficacy and safety of dornase alfa administration aerosol, intensive care hospitalized patients with COVID19-related ARDS.

The comparison of D7-D0 between the groups will be carried out using a linear regression fitted to the stratification factors.

ELIGIBILITY:
inclusion criteria

* Adult patient (age ≥ 18 years old);
* Hospitalized in intensive care ;
* Severe COVID-19 pneumonia (positive diagnosis by RT-PCR or SARS-CoV-2 antigen test on nasopharyngeal or deep respiratory specimen and/or evocative thoracic scan: frosted glass opacities, consolidation, cross-linking, thickening of interlobular septa, peripheral nodules) with ARDS criteria according to Berlin criteria (PaO2/FiO2 ≤ 300 and PEP ≥ 5).
* With respiratory assistance (intubated or NIV or ONHD) for less than 8 days;
* With an expected duration of respiratory assistance > 48 hours;
* Carrier of an arterial catheter ;
* For which 4 PaO2/FiO2 values on arterial blood over the last 24 hours are available;

Exclusion Criteria:

* Known hypersensitivity to Dornase alfa or any of the excipients;
* Pregnant or breastfeeding status;
* Patient with legal protection.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 77 (Actual)
Dates: Start 2020-04-21 (Actual); Primary Completion 2021-12-20 (Actual); Study Completion 2021-12-20 (Actual)

PRIMARY OUTCOMES:
Efficacy of intratracheal administration: occurrence of at least one grade improvement | Day 7
  The primary endpoint is the occurrence of at least one grade improvement between D0 (inclusion) and D7 in the ARDS scale severity (Berlin criteria). For instance from severe to moderate or from moderate to mild

CONTACTS AND LOCATIONS:
Overall Officials: Charles Grégoire, MD, Principal Investigator — Hôpital Fondation A de Rothschild; Julien Pottecher, MD, Study Chair — CHRU Strasbourg; Fabien Lambiotte, MD, Study Chair — CH VALENCIENNES; Serge Le Tacon, MD, Study Chair — CHR Metz-Thionville; Marie-Reine Pr Losser, Study Chair — CHRU Nancy; Pierre Kalfon, MD, Study Chair — CH Chartres; Vincent Das, MD, Study Chair — CH Montreuil; Karim Nourdine, MD, Study Chair — Hôpital Drôme Nord
Locations (1):
- Hôpital Fondation A. de Rotschhild, Paris, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Gregoire C, Di Meglio L, Le Cossec C, Ho-Tin-Noe B, Nomenjanahary MS, Guillaume J, Hamdani M, Losser MR, Lambiotte F, Le Tacon S, Cantier M, Engrand N, Yavchitz A, Trouiller P, Desilles JP, Pottecher J. Multicenter randomized trial assessing efficacy and safety of aerosolized dornase Alfa in COVID-19 ARDS. Sci Rep. 2025 Oct 22;15(1):36876. doi: 10.1038/s41598-025-20832-x. PMID 41125713
- [Derived] Desilles JP, Gregoire C, Le Cossec C, Lambert J, Mophawe O, Losser MR, Lambiotte F, Le Tacon S, Cantier M, Engrand N, Trouiller P, Pottecher J. Efficacy and safety of aerosolized intra-tracheal dornase alfa administration in patients with SARS-CoV-2-induced acute respiratory distress syndrome (ARDS): a structured summary of a study protocol for a randomised controlled trial. Trials. 2020 Jun 19;21(1):548. doi: 10.1186/s13063-020-04488-8. PMID 32560746